CLINICAL TRIAL: NCT03446833
Title: Local Field Potential (LFP) Beta Adaptive Deep Brain Stimulation (aDBS) Feasibility Study
Brief Title: LFP Beta aDBS Feasibility Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MDT17076
Record Dates: First submitted 2018-01-22; First posted 2018-02-27 (Actual); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson's Disease; Deep Brain Stimulation
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- All Subjects (Experimental): Subjects who meet the intraoperative criteria will receive The LFP Beta aDBS System.
  Interventions: Device: The LFP Beta aDBS System

INTERVENTIONS:
Device: The LFP Beta aDBS System — The LFP Beta aDBS System is intended for use in patients receiving DBS for Parkinson's Disease where LFPs may be recorded and analyzed.

SUMMARY:
The purpose of this study is to use local field potentials as control signals for adjusting DBS stimulation settings under varying patient states and to assess patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

Preoperative:

1. Subject has the ability to understand and provide written informed consent for participation in the study prior to the study-related procedures being conducted
2. Subject with levodopa-responsive PD of at least 4 years' duration, with symptoms not adequately controlled with medication, including individuals with motor complications of recent onset (from 4 months to 3 years) or with motor complications of longer-standing duration, and who are eligible for bilateral STN DBS surgery
3. Subject is ≥ 22 years of age at time of informed consent
4. Subject is a male or non-pregnant female. If female of child-bearing potential, and if sexually active, must be using, or agree to use, a medically-acceptable method of birth control as confirmed by the investigator
5. Subject has documented improvement in motor signs ON versus OFF dopaminergic medication, with a change in Unified Parkinson's Disease Rating Scale (UPDRS) Part III score of > 30% OFF to ON medication
6. Based on the opinion of the Neurosurgeon, the subject is an acceptable candidate for implant of a DBS System that includes: bilateral DBS leads targeted to the STN, extensions, and neurostimulator
7. Subject can read and understand English
8. Subject is willing and able to attend all study-required visits and complete the study procedures
9. Subject is willing and able to be awake during left and right DBS lead implant surgery and for intraoperative LFP recordings

   Intraoperative:
10. Required beta band (13 - 30 Hz) signal detected on left and right DBS leads

Exclusion Criteria

1. Subject has tremor dominant PD ≥ 2 at rest in head, upper, or lower extremities as measured on the UPDRS Part III Question 20
2. Subject requires diathermy, transcranial magnetic stimulation (TMS), or electroconvulsive therapy (ECT)
3. Subject has a history of prior intracranial surgery (eg, DBS, lesioning, previous surgical ablation)
4. Subject is unable to undergo Magnetic Resonance Imaging (MRI) of the head for planning the surgical DBS lead implants
5. Based on the opinion of the Neurosurgeon, the subject has a clinically significant structural abnormality(ies) of the brain that would jeopardize subject safety during the DBS lead implant, conduct of the study, or confound the subject's assessments
6. Subject has a metallic implant in the head, (eg, aneurysm clip, cochlear implant)
7. Subject has a major comorbidity increasing the risk of surgery (eg, prior stroke, severe diabetes, severe hypertension, immunocompromised, seizure disorder, active infection, need for chronic anticoagulation other than aspirin)
8. Subject has a neurocognitive impairment which exceeds the criteria for PD mild cognitive impairment (PD-MCI) as determined from the center's clinical neuropsychological evaluation prior to DBS for PD
9. Subject has, or plans to obtain, an implanted electrical stimulation medical device anywhere in the body (eg, cardiac pacemaker, defibrillator, spinal cord stimulator)
10. Subject has, or plans to obtain, an implanted medication pump (eg, DUOPATM infusion pump) and/or portable infusion pump
11. Based on the opinion of the investigator, the subject has an abnormal neurological examination that would preclude them from study participation
12. Subject is breast feeding
13. Subject has Mattis Dementia Rating Scale-2 (DRS-2) score ≤ 130
14. Subject has Beck Depression Inventory II (BDI-II) > 25
15. Subject is currently participating, or plans to participate, in another investigational study unless written approval is provided by the Medtronic study team

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2018-09-04 (Actual); Primary Completion 2019-02-06 (Actual); Study Completion 2019-02-06 (Actual)

PRIMARY OUTCOMES:
Operational Performance: Stimulation amplitude and LFP signals | Approximately 6 months post implant
  To characterize the stimulation amplitude and LFP signals during execution of the Medtronic LFP -based aDBS adaptive algorithm. Descriptive statistics will be reported across different PD medication states and subject activities.

SECONDARY OUTCOMES:
Acute Clinical Effect: motor examination | Approximately 6 months post implant
  The UPDRS III motor exam score will be assessed. Descriptive statistics will be reported.
Acute Clinical Effect: speech | Approximately 6 months post implant
  UPDRS III item 18 will be used to score a standardized reading passage. Descriptive statistics will be reported.
Acute Clinical Effect: dyskinesia | Approximately 6 months post implant
  UPDRS IV item 33 will be used to assess dyskinesias. Descriptive statistics will be reported.

OTHER OUTCOMES:
Number of participants with adverse events and device deficiencies | Through Study Completion, an average of 4 years
  To characterize the number of participants with serious, device-related, therapy related, and/or procedure-related adverse events and all device deficiencies assess from enrollment through study completion, using MedRA coding
Number of participants with acute stimulation-induced effects | Approximately 6 months post implant
  To characterize the number of participants with acute stimulation-induced effects of the Medtronic LFP-based aDBS algorithm assessed during all study visits that the aDBS algorithm is enabled, using MedDRA coding.

CONTACTS AND LOCATIONS:
Overall Officials: aDBS Clinical Research Team, Study Director — Medtronic RTG Brain Therapies
Locations (2):
- United States (2):
  - Stanford, Palo Alto, California
  - UPMC, Pittsburgh, Pennsylvania